CLINICAL TRIAL: NCT00711152
Title: Inclusion Of a Community Health Worker in a Collaborative Diabetes Care Program Reduces Health Care Utilization (JADE)
Brief Title: Community Health Worker Reduces Care Utilization
Acronym: JADE-MOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Asia Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Juliana Chan, Chair Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRE-2007-339
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; protocol-driven structured care; web-based; joint asia diabetes evaluation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JADE with CHW (Experimental): Patients will be enrolled into JADE program and will undergo annual comprehensive assessment (CA) with personalized JADE report with additional support by the CHW.
  Interventions: Other: Protocol-driven care under JADE Program; Other: Additional support by CHW
- JADE only (Active Comparator): Patients will be enrolled into JADE program and undergo annual comprehensive assessment (CA) with personalized JADE report without additional support by the CHW.
  Interventions: Other: Protocol-driven care under JADE Program

INTERVENTIONS:
Other: Protocol-driven care under JADE Program — The JADE Program uses the state of the art of information technology to facilitate evidence-based clinical protocol by a multidisciplinary team. There is an internet on-line and computer record system to facilitate the day-to-day management of people with diabetes.
Other: Additional support by CHW — Patients will receive additional support by a trained community health worker (CHW). Guided by the personalized report with embedded decision support, the CHW will reinforce treatment adherence and self care after each clinic visit.
  Arms: JADE with CHW

SUMMARY:
1. To recruit 600 type 2 diabetic patients managed in a community setting.
2. To enrol into the Joint Asia Diabetes Evaluation (JADE) Program.
3. All patients will undergo annual comprehensive assessment (CA) at a diabetes centre with personalized JADE report (JADE) at basline. Half of the randomized patients will be managed with additional support by a trained community health worker (CHW) (JADE+CHW).
4. All patients will undergo annual comprehensive assessments for comparison of attainment of treatment targets for 3 years

DETAILED DESCRIPTION:
Several lines of evidence support protocol-driven care using a multidisciplinary approach with special focus on periodic assessments, reinforcement of compliance and attainment of treatment targets improves risk factor control and reduces morbidity and mortality in people with diabetes mellitus The Joint Asia Diabetes Evaluation (JADE) Program is an innovative project using state of the art information technology with internet on-line system to enable doctors, nurses and other medical personnel to manage people with diabetes. It provides a virtual platform to facilitate implementation of evidence-based clinical protocols and to collect, manage and analyse data to track performance for quality assurance and improvement purposes. The JADE Program incorporates validated risk equations developed by the CUHK Diabetes Care & Research Group to stratify patients into various risk clusters for recommendation into different care protocols. This information can be relayed to people with diabetes in an interactive manner, in the form of charts and time trends, to motivate changes in behaviour and to attain treatment targets.

In this implementation project, we aim to recruit 600 type 2 diabetic patients managed in a community setting. With written informed consent, these patients will be invited to enrol into the JADE Program. All patients will undergo annual comprehensive assessment (CA) at a diabetes centre with personalized JADE report (JADE) for 3 years. Half of the patients will be managed according to the JADE protocol implemented with additional support by a trained CHW (JADE+CHW). Guided by the personalized report with embedded decision support, the CHW will reinforce treatment adherence and self care after each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of type 2 diabetes, aged 18 years or above, attending the Hospital Authority Ma On Shan Family Medicine Clinic in New Territory East Cluster
2. Type 2 diabetes is defined as follows:

   * Known history of type 2 diabetes with treatment such as lifestyle modification and/or anti-diabetic drugs for 6 months or more.
   * WHO diagnostic criteria (2 abnormal results in asymptomatic subjects or 1 abnormal result in subjects with symptoms or diabetic complications:

     * Fasting plasma glucose (PG) 7.0 mmol/L or above
     * Random PG 11.1 mmol/L or above
     * Post 75 g oral glucose tolerance test (OGTT) 2-hour PG 11.1 mmol/L or above

Exclusion Criteria:

Type 1 diabetes defined as history of ketosis [acute symptoms with heavy ketonuria (>3+) or ketoacidosis] or heavy ketonuria (>3+) or continuous requirement of insulin treatment within one year of diagnosis and thereafter.

1. Patients with terminal malignancy or other life-threatening diseases with less than 6-month expected survival
2. Telephone contact not available
3. Patients with a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2008-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin level | 3 years

SECONDARY OUTCOMES:
Cardio-metabolic control | 3 years
Number of emergency visits | 3 years
Hospitalizations with total length of stay | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Diabetes Foundation, Hong Kong, Hong Kong

REFERENCES:
- See also: Works of the Asia Diabetes Foundation — http://www.adf.org.hk